CLINICAL TRIAL: NCT04326712
Title: The Effect of Different Measurement-manufacturing Techniques on Stump and Soles Load Distribution in Transtibial Knee Prostheses
Brief Title: The Effect of Different Measurement-manufacturing Techniques on Load Distribution in Amputees
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2019.359
Record Dates: First submitted 2020-03-25; First posted 2020-03-30 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2019-04

CONDITIONS: Transtibial Amputee; Loading; Conventional; 3D
Keywords: amputee, loading, 3D

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Unilateral transtibial amputees using conventinional manufactured socket
  Interventions: Other: conventional manufactured socket
- Group 2: Unilateral transtibial amputees using 3D manufactured socket
  Interventions: Other: 3D manufactured socket

INTERVENTIONS:
Other: conventional manufactured socket — Presssure disturubition will be measured in conventional manufactured socket during walking and stairing up and down activities in unilateral transtibial amputees
  Groups: Group 1
Other: 3D manufactured socket — Presssure disturubition will be measured in 3D manufactured socket during walking and stairing up and down activities in unilateral transtibial amputees
  Groups: Group 2

SUMMARY:
Alignment of the prosthesis with the stump is performed through the socket. Good socket stump fit provides near-normal posture and weight-transfer pattern. It also ensures that the walk is painless and low-energy. Recently, studies have been carried out to use 3D printers in socket production. 3D method is accepted as an effective and reliable method in prosthetic socket production. The purpose of this study is to compare the pressures distrubution in the sockets produced by conventional and 3D scanners and printers in the transtibial amputee.

ELIGIBILITY:
Inclusion Criteria:

* Being unilateral transtibial amputation
* To have enough perception level to understand and apply commands

Exclusion Criteria:

* To have orthopedic, neurological, etc. disorder other than amputation that will affect posture or gait
* The presence of pain that will affect the posture or walking pattern
* Wound / tenderness on the stump
* Visual impairment that will affect the posture or gait pattern
* Use of any assistive device (walking stick, canary, etc.) during walking

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Unilateral transtibial amputees
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-09-06 (Actual); Primary Completion 2020-04-10 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Measurement of load distrubution on stump in conventional manufactured socket | Change from load distrubution (mmHg/N/Kg) on stump will be measured with F-socket film sensories during walking
  Load distrubution (mmHg/N/Kg) on stump will be measured with F-socket film sensories during walking.
Measurement of load distrubution on stump in 3D manufactured socket | Change from load distrubution (mmHg/N/Kg) on stump will be measured with F-socket film sensories during walking
  Load distrubution (mmHg/N/Kg) on stump will be measured with F-socket sensories during walking.
Measurement of load distrubution on stump in conventional manufactured socket | Change from load distrubution (mmHg/N/Kg) on stump will be measured with F-socket film sensories during climbing up and down stairs.
  Load distrubution (mmHg/N/Kg) on stump will be measured with F-socket film sensories during climbing up and down stairs.
Measurement of load distrubution on stump in 3D-manufactured socket | Change from load distrubution (mmHg/N/Kg) on stump will be measured with F-socket film sensories during climbing up and down stairs
  Load distrubution (mmHg/N/Kg) on stump will be measured with F-socket film sensories during climbing up and down stairs
Measurement of sole load distrubution (mmHg/N/Kg) in conventional manufactured socket | Change from sole load distrubution (mmHg/N/Kg) will be measured with F-socket film sensories during walking
  Sole load distrubution (mmHg/N/Kg) will be measured with F-scan sensories during walking
Measurement of sole load distrubution (mmHg/N/Kg) in 3D-manufactured socket | Change from sole load distrubution (mmHg/N/Kg) will be measured with F-socket film sensories during walking
  Sole load distrubution (mmHg/N/Kg) will be measured with F-scan sensories during walking
Measurement of sole load distrubution (mmHg/N/Kg) in conventional manufactured socket | Change from sole load distrubution (mmHg/N/Kg) will be measured with F-socket film sensories during climbing up and down stairs
  Sole load distrubution (mmHg/N/Kg) will be measured with F-scan sensories during climbing up and down stairs
Measurement of sole load distrubution (mmHg/N/Kg) in 3D-manufactured socket | Change from sole load distrubution (mmHg/N/Kg) will be measured with F-socket film sensories during climbing up and down stairs
  Sole load distrubution (mmHg/N/Kg) will be measured with F-scan sensories during climbing up and down stairs

CONTACTS AND LOCATIONS:
Overall Officials: yasar tatar, Study Director — Marmara University
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dou P, Jia X, Suo S, Wang R, Zhang M. Pressure distribution at the stump/socket interface in transtibial amputees during walking on stairs, slope and non-flat road. Clin Biomech (Bristol). 2006 Dec;21(10):1067-73. doi: 10.1016/j.clinbiomech.2006.06.004. Epub 2006 Aug 17. PMID 16919376
- [Background] Jia X, Suo S, Meng F, Wang R. Effects of alignment on interface pressure for transtibial amputee during walking. Disabil Rehabil Assist Technol. 2008 Nov;3(6):339-43. doi: 10.1080/17483100802044634. PMID 19127605
- [Background] Xiaohong J, Xiaobing L, Peng D, Ming Z. The Influence of Dynamic Trans-tibial Prosthetic Alignment on Standing Plantar Foot Pressure. Conf Proc IEEE Eng Med Biol Soc. 2005;2005:6916-8. doi: 10.1109/IEMBS.2005.1616096. PMID 17281865
- [Background] Lee VS, Solomonidis SE, Spence WD. Stump-socket interface pressure as an aid to socket design in prostheses for trans-femoral amputees--a preliminary study. Proc Inst Mech Eng H. 1997;211(2):167-80. doi: 10.1243/0954411971534287. PMID 9184457